CLINICAL TRIAL: NCT01255553
Title: Image Guided Partial Breast Irradiation (PBL) In A Low-Risk Population Screened With Magnetic Resonance Imaging (MRI)
Brief Title: Partial Breast Irradiation in a Low-risk Population Screened With MRI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients enrolled.
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-025-A
Record Dates: First submitted 2010-11-22; First posted 2010-12-07 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Partial Breast Irradiation — Partial breast irradiation will be administered using a 3D conformal external beam RT technique. Two fractions of 38.5 Gy separated by at least 6 hours will be given on 5 treatment days over a period of 5 to 10 days.

SUMMARY:
This is a pilot study to determine if partial breast irradiation (PBI) limited to the region of the tumor bed following lumpectomy in patients screened with MRI provides historically similar rates of local failure, limited acute skin toxicity, late complications and cosmetic outcome when compared to patients treated with standard 3D-CRT to the whole breast.

ELIGIBILITY:
Inclusion Criteria:

* Stage 0 or I breast carcinoma
* 40 years or older
* Post menopausal
* Lumpectomy with clear margins (>2mm)
* Patients with invasive disease must have undergone an axillary staging by axillary dissection (with a minimum of 6 axillary nodes) or sentinal node biopsy
* Gross disease must be unifocal with pathological tumor size 2cm or less
* Target lumpectomy cavity must be clearly marked with surgical clips (the target lumpectomy cavity/whole breast reference volume must be <=30% based on the postoperative imaging)
* Bilateral MRI of the breasts within previous 6 months of radiation therapy (RT) planning
* If patient is eligible based on postoperative imaging, partial breast irradiation (PBI) is judged to be technically deliverable
* Patients with a history of malignancies are eligible if they have stable disease as determined by their attending oncologist
* Patient must have signed the consent form

Exclusion Criteria:

* Men are not eligible
* Patients with Stage II, II, or IV breast cancer
* Pre- or peri-menopausal patients
* Patients with positive lymph nodes
* Patients with suspicious microcalcifications, densities, or palpable abnormalities unless biopsied and found to be benign
* Patients with multifocal, multicentric, or bilateral breast cancer
* Surgical margins that cannot be microscopically assessed or are positive at pathological evaluation
* Patients with a history of breast cancer
* Clear delineation of the extent of the target lumpectomy cavity is not possible
* Breast implants (patients who have had implants removed are eligible)
* Prior breast or thoracic RT for any condition

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Rates of toxicity (breast edema/pain, hyperpigmentation, erythema) for patients receiving partial breast irradiation (PBI) compared to historical rates of toxicity of patients receiving whole breast irradiation (WBI) | During radiation therapy (5-10 days)
Rates of toxicity (breast edema/pain, hyperpigmentation, erythema) for patients receiving PBI compared to historical rates of toxicity of patients receiving WBI | Post therapy (until death)

SECONDARY OUTCOMES:
Survival Rates | 5 years
Cosmetic outcomes of breast PBI | 3 years
  Comparison of cosmetic results (appearance, size, shape, texture, scaring) of breast treated with PBI to untreated breast.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Chmura, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States